CLINICAL TRIAL: NCT01803594
Title: Postprandial Modulation of HDL Metabolism
Brief Title: Feeding Trial to Determine How Combinations of Different Dietary Bioactive Ingredients Influence High Density Lipoprotein (HDL) Metabolism
Acronym: HDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 264254
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Lutein; Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Shake (Placebo Comparator): Each shake delivers 30% of each participant's calculated energy expenditure and provides 45% energy as fat, 40% energy as carbohydrate and 15% energy as protein. The shake contains whipping cream, frozen fruit, glucose polymer, and protein powder.
  Interventions: Other: Control
- PC700, Krill Oil, and Lutein (Active Comparator): Each shake delivers 30% of each participant's calculated energy expenditure and provides 45% energy as fat, 40% energy as carbohydrate and 15% energy as protein. The shake contains whipping cream, frozen fruit, glucose polymer, and protein powder. Fifty percent of the fat is made up of PC700. Additionally, 3.0g Krill oil and 40mg of lutein capsules are swallowed with water.
  Neptune Krill Oil capsules (Nutrigold); Lutein capsules (Jarrow Formulas); PC700 = dairy lipids (Fonterra brand)
  Interventions: Dietary Supplement: Krill Oil; Dietary Supplement: Lutein; Dietary Supplement: Dairy phospholipids
- PC700, Krill Oil, Lutein, and Niacin (Active Comparator): Each shake delivers 30% of each participant's calculated energy expenditure and provides 45% energy as fat, 40% energy as carbohydrate and 15% energy as protein. The shake contains whipping cream, frozen fruit, glucose polymer, and protein powder. Fifty percent of the fat is made up of PC700. Additionally, 3.0g Krill oil and 40mg of lutein capsules are swallowed with water. Nicotinic acid was added to each shake prior to consumption at a doses 5mg/kg of body weight.
  Neptune Krill Oil capsules (Nutrigold); Lutein capsules (Jarrow Formulas); PC700 (Fonterra); Nicotinic acid (Natures Way)
  Interventions: Dietary Supplement: Krill Oil; Dietary Supplement: Lutein; Dietary Supplement: Nicotinic acid; Dietary Supplement: Dairy phospholipids

INTERVENTIONS:
Dietary Supplement: Krill Oil — Neptune Krill Oil Gold
  Arms: PC700, Krill Oil, Lutein, and Niacin; PC700, Krill Oil, and Lutein
Dietary Supplement: Lutein — Jarrow Formulas
  Arms: PC700, Krill Oil, Lutein, and Niacin; PC700, Krill Oil, and Lutein
Dietary Supplement: Nicotinic acid — Natures Way
  Arms: PC700, Krill Oil, Lutein, and Niacin
Dietary Supplement: Dairy phospholipids — PC700 manufactured by Fonterra
  Arms: PC700, Krill Oil, Lutein, and Niacin; PC700, Krill Oil, and Lutein
Other: Control — Control shake without dietary supplements
  Arms: Control Shake

SUMMARY:
This study involves measuring subject's blood lipid responses after they consume a mixture of dietary fats of marine and dairy origin and vitamin supplements mixed into a milkshake, on three separate days. The investigators hope to learn more about how different food ingredients influence the metabolism HDL in individuals with low blood levels of HDL cholesterol.

DETAILED DESCRIPTION:
This study a partial randomized crossover study designed to determine how consumption of bioactive dietary ingredients in various combinations on three separate test days influences postprandial lipoprotein metabolism in participants with low circulating HDL-cholesterol.

The dietary ingredients include:

Dairy phospholipids(PC700); krill oil (K); lutein (L); and Niacin

Eligible participants will arrive to the University of California Davis (UC Davis), Ragle Human Nutrition Center on the morning of each test day after a 10-12-hr overnight fast. Upon arrival participants will fill out a questionnaire about their dietary and medication intakes and physical activity for the past 72 hours to ensure compliance. Compliant participants' weight and blood pressure will be measured and a fasting blood draw will be taken before participants consume their test meal in the form of a milkshake (control, PC700KL, PC700KL + Niacin). On each test day, participants will be given only this meal and provided with ample supply of bottled water.

Participants will only consume this test meal and water freely for the duration of the test day. Blood will be drawn serially at 2 and 4 hours postprandially. Participants will also be asked to provide 3 urine samples throughout the study: before and 2, and 4 hours after consumption of the milkshake. Participants will be tested on two additional separate test days after the first day separated by a two-week washout. The first two test days will be randomized, however the third test day will always contain niacin in order to require participants remain at Ragle for the first two hours of the study to monitor niacin flushing reactions. Participants have the option of participating in two out of three of the test days if they wish to exclude themselves from the niacin test day.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Plasma HDL cholesterol (Less than 50 mg/dL)

Exclusion Criteria:

* History of gastrointestinal disorders like Crohns disease, colitis, irritable bowel syndrome
* History of cardiovascular events: stroke, heart attack, cardiac arrhythmia
* History of peptic ulcers, gastritis
* History of gout
* History of being under care of any psychiatric conditions (schizophrenia and depression associated with response to niacin)
* Cancer
* Type 1 or 2 diabetes
* Known presence of significant metabolic disease which could impact results of study (hepatic, renal disease)
* Low blood pressure (defined as 3 consecutive readings below 100/60 mmHg at screening)
* Self report skin sensitivities; self report to rash easily
* Self report to hot flashes currently experience due to menopause
* Hypersensitivity to niacin
* Muscle disorders such as myasthenia gravis
* Pending surgery within the next 3 months
* Known allergy to study food (shellfish, fish, nut, soy)
* Known intolerance to study food (lactose intolerance)
* More than 1 serving of fish per week
* Intake of anti-inflammatory supplemental fish, krill, borage, flax, and primrose seed oils within the last 12 weeks
* Intake of dietary supplements consisting of concentrated soy isoflavones, resveratrol, other dietary polyphenols identified as modulators of lipids within the last 12 weeks
* Intake of more than 20 mg of lutein and zeaxanthin per week
* Intake of nicotinic acid (niacin) within the last 12 weeks
* Intake of anti-coagulants, blood pressure or heart medications within the last 12 weeks
* Plan to become pregnant in next 6 months
* Recent initiation (past 4 weeks) of exercise program
* Use of tobacco products
* Excessive alcohol consumption (2 drinks/day for men and 1 drink/day for women)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2013-01-02 (Actual); Study Completion 2015-03-13 (Actual)

PRIMARY OUTCOMES:
Plasma lipoprotein profile | 0, 2, 4 hour postprandial
  Plasma lipoprotein size distribution and concentration will be measured by nuclear magnetic resonance (NMR)

SECONDARY OUTCOMES:
Plasma HDL proteome | 0, 2, 4 hours postprandial
  HDL particles isolated by ultracentrifugation will be characterized for their proteomics profile measured by mass spectrometry.
Urinary metabolomics | 0, 2, 4 hours
  Urinary metabolites will be measured by NMR spectroscopy.
Red blood cell functionality | 0, 2, 4 hours postprandially
  Red blood cells isolated from whole blood will be measured for sheer stress using an in-vitro microfluidic assay.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer T Smilowitz, PhD, Principal Investigator — University of California, Davis; J. Bruce German, PhD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis, Ragle Human Nutrition Center, Davis, California, United States

REFERENCES:
- [Background] Dalbeth N, Gracey E, Pool B, Callon K, McQueen FM, Cornish J, MacGibbon A, Palmano K. Identification of dairy fractions with anti-inflammatory properties in models of acute gout. Ann Rheum Dis. 2010 Apr;69(4):766-9. doi: 10.1136/ard.2009.113290. Epub 2009 Aug 26. PMID 19713204
- [Background] Snow DR, Ward RE, Olsen A, Jimenez-Flores R, Hintze KJ. Membrane-rich milk fat diet provides protection against gastrointestinal leakiness in mice treated with lipopolysaccharide. J Dairy Sci. 2011 May;94(5):2201-12. doi: 10.3168/jds.2010-3886. PMID 21524510
- [Background] Mozaffarian D, Rimm EB, Herrington DM. Dietary fats, carbohydrate, and progression of coronary atherosclerosis in postmenopausal women. Am J Clin Nutr. 2004 Nov;80(5):1175-84. doi: 10.1093/ajcn/80.5.1175. PMID 15531663
- [Background] Tholstrup T, Vessby B, Sandstrom B. Difference in effect of myristic and stearic acid on plasma HDL cholesterol within 24 h in young men. Eur J Clin Nutr. 2003 Jun;57(6):735-42. doi: 10.1038/sj.ejcn.1601605. PMID 12792657
- [Background] Bunea R, El Farrah K, Deutsch L. Evaluation of the effects of Neptune Krill Oil on the clinical course of hyperlipidemia. Altern Med Rev. 2004 Dec;9(4):420-8. PMID 15656713
- [Background] Ribaya-Mercado JD, Blumberg JB. Lutein and zeaxanthin and their potential roles in disease prevention. J Am Coll Nutr. 2004 Dec;23(6 Suppl):567S-587S. doi: 10.1080/07315724.2004.10719427. PMID 15640510
- [Background] Kiokias S, Gordon MH. Dietary supplementation with a natural carotenoid mixture decreases oxidative stress. Eur J Clin Nutr. 2003 Sep;57(9):1135-40. doi: 10.1038/sj.ejcn.1601655. PMID 12947433